CLINICAL TRIAL: NCT04659785
Title: A Single-Arm,Single-Center, Phase Ib/II Clinical Study of Fluzoparib (SHR-3162) Combined With Apatinib as Second-Line Treatment of Patients With Extensive Stage Small Cell Lung Cancer（SCLC）
Brief Title: A Study of Fluzoparib Combined With Apatinib as Second-Line Treatment of Patients With Extensive Stage Small Cell Lung Cancer（FA-ES-SCLC）
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-SCLC-2nd-IIT-SHR3162-APA
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Small Cell Lung Cancer Extensive Stage
Keywords: Fluzoparib; Apatinib; Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — fluzoparib; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzoparib + Apatinib (Experimental): Fluzoparib and apatinib will be administered continuously and orally in combination, 28 days per cycle, until disease progression or unacceptable toxicity.
  Interventions: Drug: Fluzoparib; Drug: Apatinib

INTERVENTIONS:
Drug: Fluzoparib — Take Fluzoparib orally（either at 50,100mg bid）until disease progression or appearance of unbearable toxicity
  Other Names: SHR3162; HS10160
Drug: Apatinib — Take apatinib orally (either at 375mg、500mg、750mg qd）until disease progression or appearance of unbearable toxicity
  Other Names: Apatinib mesylate

SUMMARY:
This open-label, dose finding phase Ib trial studies the tolerability and the best dose of fluzoparib in combination with apatinib and to see how well these two drugs work together as second-line treatment of patients with extensive stage small cell lung cancer. The safety and efficacy of fluzoparib in combination with apatinib will be explored. Both dose escalation and dose expansion parts are included in this study.

DETAILED DESCRIPTION:
The degree of malignancy of small cell lung cancer is extremely high. About 60% to 70% of patients are diagnosed as extensive. The median survival time of the disease is only 9 to 10 months, and the 2-year survival rate is less than 10%. Fluzoparib is an oral potent, selective poly-ADP ribose polymerase-1 (PARP-1) and PARP-2 inhibitor. Apatinib is an oral selective vascular endothelial growth factor receptor (VEGFR) inhibitor.This open-label, dose finding phase Ib trial studies the tolerability and the best dose of fluzoparib in combination with apatinib as second-line treatment of patients with extensive stage small cell lung cancer. The safety and efficacy of fluzoparib in combination with apatinib will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Extensive Stage Small Cell Lung Cancer diagnosed by pathology (histology or cytology) (according to WHO classification in 2015);
2. Failure of first-line treatment；
3. Age 18-70 years old;
4. ≤21 days before the first study drug, CT or MRI scan, at least one target lesion without previous radiotherapy as defined by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1);
5. PS score: 0-2; the expected survival time ≥ 12 weeks;
6. No anti-angiogenesis drugs or PARP inhibitors have been used in previous treatments;
7. All acute toxic reactions caused by previous anti-tumor treatments or surgical operations were relieved before the screening period 0-1 grade (according to NCI CTCAE 5.0 judgment) or to the level specified by the inclusion/exclusion criteria (hair loss and other researchers believe that the subjects are not Except for toxicity that poses a safety risk);
8. No blood transfusion or blood products, no correction with G-CSF and other hematopoietic stimulating factors within 14 days before the first administration. First research before investigating drugs, laboratory test values meet the following conditions:

   1. Blood routine: white blood cell count (WBC) ≥3.0 × 109/L; absolute neutrophil count (ANC) ≥1.5 × 109/L; Platelet (PLT) ≥100 × 109/L; Hemoglobin content (HGB) ≥9.0 g/dL;
   2. Liver function: Aspartate aminotransferase (AST) ≤2.5 x ULN in subjects without liver metastasis, alanine liver aminotransferase (ALT) ≤2.5 x ULN; ALT and AST in subjects with liver metastases <5 x ULN; Serum total bilirubin (TBIL) ≤1.5 x ULN (except Gilbert syndrome total bilirubin <3.0 mg/dL); Albumin (ALB) ≥3 g/dL;
   3. Renal function: serum creatinine ≤1.5 x ULN or creatinine clearance CrCl≥40 mL/minute;
   4. Coagulation function: International normalized ratio (INR) ≤ 1.5, activated partial thromboplastin time (APTT) ≤ 1.5 x ULN;
   5. Others: Lipase ≤ 1.5 x ULN, if lipase> 1.5 x ULN but no clinical or imaging confirmed pancreatitis can be included; amylase ≤ 1.5 x ULN, if amylase> 1.5 x ULN but no clinical or imaging confirmed pancreatitis can be included in the group. Alkaline phosphatase (ALP)≤2.5ULN, subjects with bone metastases, ALP≤5ULN;
9. Non-surgically sterilized female subjects of childbearing age must have a negative serum HCG test within 3 days before the first medication, and non-lactating period. Male subjects and females of childbearing age must start the first study drug to after the last study drug 6 contraception within months;
10. Subjects voluntarily join the study, with good compliance, with safety and survival follow-up.

Exclusion Criteria:

1. Active brain metastases or meningeal metastases with clinical symptoms. Subjects with treated brain metastases need to meet the following conditions to be tested considered into the group:

   1. It is confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) that the lesion is stable since the end of treatment≥4 weeks;
   2. No need to receive systemic corticosteroids (>10mg/day prednisone or equivalent dose) treatment;
2. The third space effusion with clinical symptoms, such as pericardial effusion, pleural effusion and effusion that cannot be controlled by pumping or other treatments ascites;
3. People with symptoms of cough, hemoptysis, bloody sputum within 1 month before the first medication;
4. Minor surgery (including catheterization) was performed within 48 hours before the first study drug;
5. Other anti-tumor drugs are currently being used within 4 weeks after the last systemic cytotoxic drug treatment or radiotherapy drug treatment;
6. Currently or recently (within 30 days before enrollment) using another investigational drug or participating in another clinical study;
7. Other malignant tumors (fully treated cervical carcinoma in situ or skin squamous cell carcinoma, or controlled skin except for basal cell carcinoma);
8. Have previously received PARP inhibitors or small molecule inhibitors targeting vascular endothelial cell growth factor receptor (VEGFR) agent treatment;
9. Patients with hypertension who cannot be reduced to the normal range after treatment with antihypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
10. There are clinical symptoms or diseases of the heart that are not well controlled, such as: I. Heart failure above NYHA 2; II. Instability Stereotyped angina; III. Myocardial infarction occurred within 1 year; IV. clinically significant supraventricular or ventricular arrhythmia needs treatment or intervention; V QTc>470ms;
11. Abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5 ULN), with have a bleeding tendency or are receiving thrombolysis or anticoagulation therapy;
12. Have significant clinically significant bleeding symptoms or have a clear bleeding tendency within 3 months before signing the ICF (Information Consent Form), such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood++ and above, or suffering from vasculitis;
13. Arterial/venous thrombotic events, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc;
14. Have the following medical history within 24 weeks before signing the ICF: peptic ulcer, gastrointestinal perforation, corrosive esophagitis or gastritis, inflammation enteropathy or diverticulitis, abdominal fistula, tracheo-esophageal fistula, or intra-abdominal abscess;
15. Major surgery or severe traumatic injury, fracture or ulcer occurred within 4 weeks before treatment;
16. There are factors that significantly affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
17. Urine routine test indicates urine protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0 g;
18. The investigator judges other situations that may affect the conduct of clinical research and the judgment of research results;
19. Patients with a clear history of allergies may be potentially allergic or intolerant to Apatinib and Fluzoparib;
20. Human immunodeficiency virus (HIV) infection, active hepatitis B (hepatitis B surface antigen positive and HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody is positive and HCV-RNA is higher than the detection limit of the analytical method);
21. According to the judgment of the investigator, there is an accompanying disease (such as poorly controlled hypertension, severe diabetes, neurological or mental illness, etc.) that seriously endangers the safety of the subject, may confuse the research results, or affects the subject to complete the study Any other situation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase Ⅰb: Determination of Recommended Phase II dose (RP2D) of Escalating Dose of Fluzoparib with Apatinib | Up to 28 days after the first dose of Fluzoparib and Apatinib combination therapy
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for the dose expansion arms, based on safety, tolerability and efficacy data collected during the dose escalation portion of the study
PhaseⅠb: Incidence of Adverse Events [safety and tolerability] | From screening up to 28 days after end of treatment
  Adverse events defined according to Common Terminology for Adverse Events (CTCAE) v5.0
Phase Ⅱ: Objective Response Rate(ORR) as Assessed by the Investigator according to RECIST v1.1 | up to approximately 2 Years
  Objective Response Rate(Complete response + Partial response (CR+PR)), determined using RECIST v1.1 criteria, defined as best overall response (complete or partial response) across all assessment time points.

SECONDARY OUTCOMES:
Progression Free Survival（PFS） | Up to approximately 2 Years
  Progression Free Survival, defined as first assessment of disease progression or death, whichever is earlier.
Overall survival（OS） | Up to approximately 2 Years
  Overall survival is the time from intervention to death due to any reason or lost of follow-up
Duration of Response（DoR） | Up to approximately 2 Years
  Duration of Response, determined using RECIST v1.1 criteria.
Adverse Event Rate（AER） | Up to approximately 2 Years
  Adverse events defined according to Common Terminology for Adverse Events (CTCAE) v5.0
Biomarker Detection | Up to approximately 2 Years
  Evaluation of TP53 gene status through next-generation sequencing technology

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Wang, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality, China